CLINICAL TRIAL: NCT07166042
Title: Med-RT BG: An Interventional Trial Using Guided Meditation During Radiation Therapy for Breast and Gynecological Malignancies
Brief Title: Guided Meditation During Radiation Therapy for Breast and Gynecological Malignancies
Acronym: Med-RT BG
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCI192768
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer; Gynecologic Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided Meditation Intervention (Experimental)
  Interventions: Behavioral: 10-15 minute, Audio-Recorded Guided Mediation Practices
- Standard of Care (No Intervention)

INTERVENTIONS:
Behavioral: 10-15 minute, Audio-Recorded Guided Mediation Practices — The 5 mindfulness practices, all of which have been validated in prior research.
  Body Scan practice will consist of how to direct non-judgmental attention to different regions of the body
  The Mindful Breathing practice will consist of focused attention on the breath and metacognitive monitoring and acceptance of discursive thoughts, negative emotions, and body sensations.
  The Mindfulness of Discomfort practice will consist of instruction in how to "zoom in" to deconstruct discomfort and precisely map each feelings' spatial location, use mindful breathing to "zoom out" and broaden the field of awareness to include neglected sensory elements, and shift attention from unpleasant feelings to neutral/pleasant sensations or experiences.
  The Savoring practice will consist of instruction in identifying and amplifying pleasant memories.
  The Loving-Kindness practice will consist of instruction in cultivating feeling of warmth and compassion toward the self and others.
  Arms: Guided Meditation Intervention

SUMMARY:
The goal of this study is to assess the effect of brief mindfulness-guided meditations during radiation therapy (RT) for patients with anxiety related to RT for breast and gynecological cancers.

ELIGIBILITY:
Inclusion Criteria:

* Participant aged ≥ 18 years.
* Diagnosis of breast or gynelogical cancer.
* Eligible to receive 15-25 daily radiation therapy treatments for breast or gynelogical cancer.
* Willing to participate in either the guided meditation or standard of care control arm, regardless of treatment assignment.
* Karnofsky performance score ≥ 60 or ECOG performance score ≤ 2.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* Active suicidal ideation or active psychotic state in the opinion of the investigator.
* Patient is receiving deep inspiration breath hold treatment.
* An unstable illness that, in the opinion of the investigator, would interfere with study treatment.
* Prior radiation therapy.
* Inability to understand and/or speak the English language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in acute anxiety in participants receiving mindfulness intervention during RT compared to standard of care control conditions. | 7 weeks
  To assess the acute anxiolytic effects of a brief mindfulness intervention during radiation therapy (RT) for patients with anxiety related to RT for breast and gynecological cancers.
  Acute anxiety during RT will be measured at each treatment visit with an individual item ("How nervous, anxious or on edge do you feel right now?" scored on a 0 (not at all) to 10 (Very much). derived from the Generalized Anxiety Disorder 2-item (GAD-2) scale, measured before and after RT. The change from before to after RT will be averaged over all treatment visits.

SECONDARY OUTCOMES:
Change in anxiety in everyday life in participants receiving mindfulness intervention during RT compared to standard of care control conditions. | 7 weeks
  To assess the distal anxiolytic effects of a brief mindfulness intervention during RT for patients with anxiety related to RT for breast and gynecological cancers.
  Anxiety in everyday life will be measured using the total score of the Generalized Anxiety Disorder 2-item (GAD-2) scale prior to RT (minimum value 0, maximum value 6, score of 3 or higher considered clinical). This will be measured once a week during RT.
Change in anxiety during RT and in everyday life as measured by the modified MPoD | 7 weeks
  To determine whether the brief mindfulness intervention during RT increases patients' state mindfulness and whether the degree of changes in state mindfulness during RT predict decreases in acute anxiety and anxiety in daily life.
  Modified Metacognitive Processes of Decentering Scale (MPoD) consists of 4 items scored on a 0-10 scale, "0" meaning "Not at All" and "10" meaning "Very Much".
Change in self transcendence and the magnitude/degree of increased self transcendence will predict degree of anxiety in the course of daily life as measured by total score of the Nondual Awareness Dimensional Assessment (NADA). | 7 weeks
  To determine whether the brief mindfulness intervention during RT increases patients' self transcendence and whether the degree of changes in self-transcendence during RT predict decreases in anxiety in daily life. The NADA will ask patients to rate their feelings 15 minutes before and after treatment on a scale of 0 (not at all) to 10 (very much).

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Burt, MD, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah, United States